## Assessment by Ultrasound of the degree of venous dilatation, comparison between venodilation by Airglove™ versus Warm Water Immersion (WWI)

HLS/PSAWAHS/18/168

25th March 2019



## ASSESSMENT BY ULTRASOUND OF THE DEGREE OF VENOUS DILATION; COMPARISON BETWEEN AIRGLOVE™ AND WARM WATER IMMERSION (WWI) METHOD

## **ELAINE GARDINER**

## **CONSENT FORM**

| | | | Please ir | nitial box |
|---|---|---|---|---|
| 1. | I confirm that I have read and under<br>(version 1) for the above study and<br>questions and have had these answ | have had the opportu | | |
| 2. | I understand that my participation is any time without giving any reason affected. | • | | |
| 3. | I agree to take part in the above stu | ıdy. | | |
| 3. | I understand that information provid<br>and may be used in publications ab<br>possible to identify me from this info | out the research how | vever it will not be | ed |
| 5. | I consent to allow my basic demogration secure server. The data held on the further analysis and in comparison the Life Sciences at Glasgow Caledon | database will not be with future data, by st | identifiable. This data may be | used for |
| 6. | I understand that the results from thi possible to identify any participant | | shed however it will not be | |
| | agree that any unexpected findings permission for this. | will be reported to m | y General Practitioner. I give | |
| Name | or initials of participant | <br>Date | Signature or initials | |

| Name of person taking consent (if different from researcher) | Date | Signature |
|---|---|---|